CLINICAL TRIAL: NCT02433106
Title: The Effects of an Exercise Based Injury Prevention Programme on Neuromuscular Outcomes in Gaelic Football and Hurling Players, a Randomised Controlled Trial
Brief Title: The Effects of an Exercise Programme on Neuromuscular Outcomes in Gaelic Sport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Ulrik McCarthy Persson (Other)
Responsible Party: Sponsor-Investigator, Dr Ulrik McCarthy Persson, Dr, University College Dublin
Organization: University College Dublin (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GAA intervention
Record Dates: First submitted 2015-04-20; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Focus of Study is Effects of Neuromuscular Training
Keywords: Balance; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): GAA 15 Specific neuromuscular exercise training
  Interventions: Other: GAA 15
- Control (Active Comparator): Control Usual training
  Interventions: Other: Control

INTERVENTIONS:
Other: GAA 15 — Neuromuscular injury prevention training
  Arms: Intervention
Other: Control — Usual training
  Arms: Control

SUMMARY:
A randomized control trial examining the effects of an exercise based injury prevention programme on postural control and jump landing mechanics. Randomization of 4 teams, 2 Gaelic football and 2 hurling teams to exercise intervention and control groups. Participants are tested using Y Balance test and Landing Error Scoring System (LESS).

DETAILED DESCRIPTION:
Gaelic football and hurling, a stick and ball game, are Irish amateur games components of explosiveness with the multi-directional nature of both games, in addition to the overhead activities and the high level of contact involved; makes it a high risk of injury, especially during match-play. Recent systematic reviews found that injury prevention exercise programmes can significantly reduce the relative risk of lower extremity injuries. Several studies have successfully incorporated exercise components including balance, plyometrics, strength, neuromuscular training, running and cutting movement patterns to prevent injuries in sports such as soccer, basketball, and handball.

This study examines the effect of an injury prevention programme on 2 recognized risk factors for lower limb injury balance and jump landing mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered on Collegiate Gaelic football or hurling team, which trained at least twice per week.
* To be over the age of 18 years
* No current injuries

Exclusion Criteria:

* Injuries of the lower limb preventing training or completing the testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Y Balance test | baseline to 8-weeks
  Dynamic balance reach test

SECONDARY OUTCOMES:
Landing error scoring system | baseline to 8-weeks
  Assessment of jump landing movement pattern

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Blake, PhD, Study Director — UCD
Locations (1):
- University College Dublin, Dublin, Ireland